CLINICAL TRIAL: NCT06950515
Title: A Randomized Controlled Trial of gEneral aneStheSia vs consciOUs Sedation in Radial endobronChial Ultrasound for Peripheral Pulmonary lEsions
Brief Title: General Anesthesia vs Conscious Sedation for Radial Endobronchial Ultrasound
Acronym: RESSOURCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Marc Fortin, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2025-4122
Record Dates: First submitted 2025-02-14; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancers; Peripheral Pulmonary Nodules
Keywords: Lung cancer; Peripheral pulmonary nodules; bronchoscopy; peripheral endobronchial ultrasound; sedation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized clinical trial to compare the diagnostic yield of pEBUS under general anesthesia and conscious sedation in the context of the investigation of peripheral pulmonary lesions.
Who Masked: Outcomes Assessor
Masking Description: The pathologist will be blinded when reviewing biopsy specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conscious sedation arm (Experimental): In the conscious sedation group, the procedure will be performed through the nose or mouth at the discretion of the endoscopist. The patient will remain breathing spontaneously throughout the procedure and will be administered oxygen through a nasal cannula at an initial flow rate of 2L/min. A combination of propofol, fentanyl and midazolam boluses will be used to maintain moderate sedation. At IUCPQ-UL, fentanyl and midazolam will be used as in our routine practice. The boluses will be prescribed by a doctor experienced in conscious sedation (anesthesiologist, intensivist or pulmonologist) according to the patient's state of wakefulness assessed by the Richmond Agitation-Sedation Scale (RAS) .Centers will decide, prior to initiating recruitment locally, the drug combination used to sedate patients and they will maintain the use of the same drug combination throughout the study.
  Interventions: Procedure: Peripheral EBUS under Concious sedation
- General anesthesia arm (Experimental): In the general anesthesia group, an endotracheal tube larger than 7 will be used. The patient will be kept non-arousable to non-nociceptive stimulation (RAS = -5) by a perfusion including, at the anesthesiologist's discretion: fentanyl, sufentanyl, remifentanyl, midazolam or propofol. The sedation of this group will not be protocolized given the wide variety of practices in the participating centers, but the targeted level of sedation will be and the medication administered will be adjusted according to this target. The RAS will be evaluated every 5 minutes, or earlier if signs of arousal are present, to ensure that the intended target is maintained and adjustments to the rate of infusions as well as boluses may be made/administered by the anesthesiologist to maintain the targeted level of sedation. Patients may be paralyzed at the discretion of the anesthesiologit. The ventilatory parameters will be standardized according to the VESPA protocol
  Interventions: Procedure: Peripheral EBUS under General Anesthesia

INTERVENTIONS:
Procedure: Peripheral EBUS under Concious sedation — In the conscious sedation group, the procedure will be performed through the nose or mouth at the discretion of the endoscopist. The patient will remain breathing spontaneously throughout the procedure and will be administered oxygen through a nasal cannula at an initial flow rate of 2L/min. A combination of propofol, fentanyl and midazolam boluses will be used to maintain moderate sedation. At IUCPQ-UL, fentanyl and midazolam will be used as in our routine practice. The boluses will be prescribed by a doctor experienced in conscious sedation (anesthesiologist, intensivist or pulmonologist) according to the patient's state of wakefulness assessed by the Richmond Agitation-Sedation Scale (RAS) .Centers will decide, prior to initiating recruitment locally, the drug combination used to sedate patients and they will maintain the use of the same drug combination throughout the study
  Arms: Conscious sedation arm
Procedure: Peripheral EBUS under General Anesthesia — In the general anesthesia group, an endotracheal tube larger than 7 will be used. The patient will be kept non-arousable to non-nociceptive stimulation (RAS = -5) by a perfusion including, at the anesthesiologist's discretion: fentanyl, sufentanyl, remifentanyl, midazolam or propofol. The sedation of this group will not be protocolized given the wide variety of practices in the participating centers, but the targeted level of sedation will be and the medication administered will be adjusted according to this target. The RAS will be evaluated every 5 minutes, or earlier if signs of arousal are present, to ensure that the intended target is maintained and adjustments to the rate of infusions as well as boluses may be made/administered by the anesthesiologist to maintain the targeted level of sedation. Patients may be paralyzed at the discretion of the anesthesiologit. The ventilatory parameters will be standardized according to the VESPA protocol
  Arms: General anesthesia arm

SUMMARY:
The endoscopic investigation of lung lesions is experiencing significant growth with the increasing number of lung cancer screening programs. Peripheral endobronchial ultrasound (pEBUS) is the most widely used endoscopic technique in the investigation of peripheral pulmonary lesions (PPL). It is performed in relatively equal proportions under conscious sedation and general anesthesia by interventional pulmonologists throughout the world. Users of conscious sedation justify themselves by the fewer resources consumed and the absence of demonstration of a superior diagnostic yield of general anesthesia while users of general anesthesia claim diagnostic yield and comfort for the patient are superior with their approach. Our main objective is to compare the diagnostic yield of pEBUS under general anesthesia to that obtained under conscious sedation.

DETAILED DESCRIPTION:
This is a multicenter randomized clinical trial to compare the diagnostic yield of pEBUS under general anesthesia and conscious sedation in the context of the investigation of peripheral pulmonary lesions.

Participants will be recruited prospectively. Potential participants will be identified during the screening of procedure requisitions by the interventional pulmonology team. The participant will then be approached by the physician to obtain their consent to the procedure and the study during a first visit, which can be face-to-face, by phone or by telemedicine. During this visit, the research protocol and the risks involved will be explained to the participant by the physician to obtain their free and informed consent for both. After verifying eligibility criteria and obtaining consent, participants will be included in the study and randomized. Participants will be randomized to the type of sedation for the procedure (general anesthesia or conscious sedation) and the procedure can, then, be scheduled with the sedation mode assigned during randomization. During a second visit, which may take place on the same day as the first, the participant will undergo pEBUS under conscious sedation or general anesthesia depending on the group to which he was randomized. Prior to discharge, the participant's comfort questionnaires will be administered. One month after the procedure, the research team will consult the participant's medical record to review the results of the samples taken during the examination and to ensure that the participant have not suffered any late complications following the procedure. The patient will be instructed to contact the research team again if they believe they have had a late complication. The record will subsequently be reviewed at 1 and 2 years if the procedure is not diagnostic to validate the final clinical diagnosis of the treating team. Communication of the results and further treatment of the patient will be the responsibility of the referring physician or his team and not that of the research team.

In both groups, a MP190 or P180/190 bronchoscope (Olympus, Tokyo, Japan) and a UM-S20-17S or 20R-3 radial EBUS probe (Olympus, Tokyo, Japan) will be used. A guidesheath will be used when performing pEBUS procedures with a P180/190 bronchoscope but not when using a MP190. Each center will determine before beginning recruitment for the study whether if it will use a P180/190 with guidesheath or a MP190 without guidesheath. This center must systematically use the same type of bronchoscope, for all participants recruited according to their predetermined conduct. Minimally, a wash, forceps and a brush will be performed to sample the lesion. Forceps biopsies will be taken until five macroscopically visible specimens are obtained, up to a maximum of 8 attempts. A single brushing as well as a cytological bronchoalveolar washing, of at least 50ml, will be carried out. At the discretion of the center, a peripheral needle for fine aspiration may also be used (eg. Periview, Olympus, Tokyo, Japan). If used, a minimum of 3 passes will be performed, but additional passes are permitted at the discretion of the endoscopist and depending on the material obtained macroscopically. Each center will determine before beginning recruitment for the study whether or not it will use a fine needle technique. This center must systematically use it or not, for all participants recruited according to their predetermined conduct.

A 1.1mm cryoprobe (Erbe, Tuebingen, Germany) can also be used at the discretion of the endoscopist. The cryoprobe will only be used in the general anesthesia group as the risk of hemorrhage with this technique is prohibitive in the non-intubated patient. Cryobiopsies do not have to be performed or not performed in all participants in a center, in contrast to fine needle aspiration, and can be used at the discretion of the bronchoscopist. The sequence of samples will be at the discretion of the endoscopist. No rapid on-site cytology analysis will be performed in either group.

Randomization will be carried out at the end of the first visit to allow the logistical organization of the second visit, which includes the intervention. A 1:1 randomization, stratified for center and the presence of a bronchus sign will be performed. A bronchus sign will be defined by the presence of a bronchus leading directly to the lesion. Randomization will be centralized using the RedCapMD computer platform including a computer-generated randomization table by a consultant statistician. Participating centers will not have access to the randomization table. The participant and the medical team performing the intervention cannot realistically be blinded to the group to which the participant was randomized, but the primary outcome will depend on the impression of the pathologist and physician reviewing the chart who will be blinded to the randomization group. The pathologist will also be blinded to the cryoprobe biopsies when reviewing other biopsies of the same patient (forceps, brush, fine needle and wash) to prevent contamination of his final diagnosis for the other biopsies by the cryoprobe biopsy. The cryoprobe biopsy will be reviewed by a second pathologist or the same pathologist after recording is impression for the other biopsies. At no time before the end of the study can the blinding be lifted for the pathologist or physician reviewing the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ability to consent
* Peripheral lung lesion less than 5cm in average diameter on axial CT images (A lung lesion will be considered peripheral if it is located beyond the origin of the subsegmental bronchi and presumed not to be visible endoscopically in white light during the evaluation of the CT scan by an interventional pulmonologist.)
* Lesion deemed accessible by pEBUS by an experienced interventional pulmonologist
* Decision by the medical team and the patient to use pEBUS as a diagnostic modality for the lung lesion

Exclusion Criteria:

* Planned use of electromagnetic navigation, augmented fluoroscopy or robotic bronchoscopy in addition to pEBUS. The use of virtual bronchoscopy planning is permitted
* Presence of suspicious lymph nodes (size ≥ 10mm and/or moderate or greater hypermetabolism) on imaging which are accessible by l-EBUS and for which rapid on-site cytological analysis will be used
* Contraindication to bronchoscopy or biopsies such as an unstable medical condition or uncorrected coagulopathy
* Current pregnancy
* Lack of free and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of pEBUS under general anesthesia and conscious sedation | At recruitment completion (expected time 2 years)
  The diagnostic yield of pEBUS according to a strict definition, a procedure being defined as diagnostic if it allows a specific benign or malignant diagnosis using the samples obtained. Non-specific findings not allowing a precise diagnosis and accompanied by a follow-up evolution consistent with the findings (e.g.: non-specific inflammation followed by spontaneous resolution of the lesion) will not be considered diagnostic. Cryobiopies will be excluded from the primary outcome as they cannot be safely performed under conscious sedation. We do not primarly aim to evaluate the added value of cryobiopsy but to compare two modalities of sedation.
  The comparison between the diagnostic yields for the two types of sedation will be made with a χ2 test, if the distribution of the data is normal

SECONDARY OUTCOMES:
Diagnostic yield of pEBUS | At recruitment completion (expected time 2 years)
  The diagnostic yield of pEBUS according to a strict definition with inclusion of cryobiopsy results.
  The comparison of the variables will be carried out with a χ2 test
Diagnostic yield of pEBUS | At recruitment completion (expected time 2 years)
  The diagnostic yield of pEBUS according to a strict definition, with and without inclusion of cryobiopsy results, amongst lesions under and over 20mm of average diameter.
  The comparison of the variables will be carried out with a χ2 test
Diagnostic yield of pEBUS | At recruitment completion (expected time 2 years)
  The diagnostic yield of pEBUS according to a liberal definition, a procedure being defined as diagnostic if it allows a specific benign or malignant diagnosis or if it demonstrates non-specific inflammation and that during follow-up a precise benign diagnosis is established or that the lesion regresses on serial imaging. This analysis will be performed with and without inclusion of cryobiopsies.
  The comparison of the variables will be carried out with a χ2 test
Duration of the procedure | Assessment will begin with the start of the procedure (bronchoscope insertion) and end at procedure completion (bronchoscope removal)
  The duration of the procedure from insertion of the bronchoscope to its removal, excluding the time spent on l-EBUS if applicable
Duration of the procedure | Assessment will begin when the participant enters the procedure room and end when he leaves it. Result will be recorded when the patient leaves the procedure room.
  The duration of the procedure from patient's procedure room entry to his departure from the procedure room.
Recovery duration | Assessment will begin when the participant leaves the procedure room and end when he is discharged from the recovery room. Result will be recorded when the patient is discharged from the recovery room.
  The duration of post-procedure recovery before reaching the criteria for discharge (PADS ≥ 9 and adequate oxygen saturation)
Participant Comfort | Questionnaires will be administered once the patient is ready for discharge from the recovery room
  Comfort during the examination according to the patient measured by visual analogue scale (in millimeters, from 0 to 100mm, with 0mm corresponding to no discomfort and 100mm to severe discomfort) and two Likert scales of memory of the procedure (absolutely no memory, no specific details, a few details, most of the details, all the details) and willingness to repeat the examination if medically required (definitely not, probably not, uncertain, probably, definitily)
Adverse event rates | At recruitment completion (expected time 2 years)
  The rate of adverse events and serious adverse events of pEBUS under general anesthesia versus conscious sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided